CLINICAL TRIAL: NCT06118112
Title: Living With Long COVID: LONGCOVID-EXPERIENCE Qualitative Study
Brief Title: Living With Long COVID: LONGCOVID-EXPERIENCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Principal Investigator, Anna Selva, Co-principal investigator, Corporacion Parc Tauli
Other Study IDs: LONGCOVID EXPERIENCE
Record Dates: First submitted 2023-09-15; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Long COVID; Experience, Life
Keywords: Post-Acute COVID-19 Syndrome; patient experience; qualitative research
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with- long-covid: Women and men diagnosed with persistent COVID according to WHO (World HEalth Organization) criteria: persistent symptoms three months after the acute manifestations of COVID-19 and lasting at least two months and cannot be explained by an alternative diagnosis.

SUMMARY:
Background: One in ten people infected with COVID-19 presents persistent COVID, which consists of the presence of symptoms three months after the acute manifestations of COVID-19 and their persistence for at least two months, without being explained by an alternative diagnosis. The characteristics and clinical approach to persistent COVID syndrome are fairly well known, but not what the experience of people with persistent COVID is in relation to their daily life, their work life, and their experience with the healthcare received. Objective: to understand the experience of patients with persistent COVID in relation to the disease, the health care received and re-entry into the world of work

Methods: Qualitative, descriptive, phenomenological study, based on individual interviews. The study protocol will be registered in Clinicaltrials.gov. People with persistent COVID treated at the Parc Taulí Hospital will be included. Sampling will be by convenience, purposive and snowball and the sample size will be determined by data saturation. Semi-structured individual or group interviews will be conducted and the data will be analyzed following a reflective thematic analysis (Brawn and Clarke). The preliminary report will be triangulated with some participants and with the results obtained from a scoping review carried out by the research team.

ELIGIBILITY:
Inclusion Criteria:

* women and men diagnosed with persistent COVID between March '20 to the present according to WHO criteria (persistent symptoms three months after the acute manifestations of COVID-19 and lasting at least two months and cannot be explained by an alternative diagnosis).
* treated at the Parc Taulí Hospital
* from 18 to 65 years

Exclusion Criteria:

-people who do not understand or can communicate in Catalan or Spanish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the Parc Taulí Hospital Universitari, a hospital with a reference population of 400,000 urban people and 4,500 workers.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Experience of the disease | Up to three years
  How is living with LongCOVID. Assessed through semi-structured interviews.
Experience with healthcare received | Up to three years
  How is the experience of patients with the healthcare received for their condition. Assessed through semi-structured interviews.
Experience with return to work | Up to three years
  What were the barriers and facilitators for returning to work after the disease. Assessed through semi-structures interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Selva, MD, MPH, PhD, Principal Investigator — Parc Taulí, Hospital Universitari- I3PT; Juan Leiva, PhD, Study Director — Universitat Autònoma Barcelona; Pilar Peña, MD, Principal Investigator — Parc Taulí, Hospital Universitari- I3PT
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No